CLINICAL TRIAL: NCT03703128
Title: Psychological Autopsy Study: A Case-control Research Into 45-60 Year Old Suicide Victims in Flanders, Belgium
Brief Title: Suicide in People Aged 45-60: A Case-control Psychological Autopsy Study
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: Flemish Ministry of Welfare, Public Health, and Family, Belgium (Unknown)
Responsible Party: Sponsor
Other Study IDs: B670201836751
Record Dates: First submitted 2018-09-27; First posted 2018-10-11 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Suicide
Keywords: psychological autopsy; prevention
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Informants of suicide victims: Partners, children, parents, siblings, other relatives, peers or other informants of adults (aged 45-60 years) who received a definitive verdict of suicide in the Dutch-speaking part of Belgium (Flanders). The suicide should have taken place more than 3 months ago and less than 5 years ago.
- Control group: Informants i.e., partners, children, parents, siblings, other relatives, peers or other informants of adults (aged 45-60 years) who have mental health problems.

SUMMARY:
The purpose of this study is to learn about the possible causes of the negative trend in suicide rates in both males and females aged 45-60 in Flanders, Belgium. This will be carried out using a psychological autopsy study.

DETAILED DESCRIPTION:
A case-control psychological autopsy study will be carried out to identify what risk factors are related to suicide in people aged 45-60. People close to the person who died by suicide (next of kin or close friends) will be interviewed. To increase the validity of our findings, a control group will also be interviewed. The control group will be someone who is very close to someone with mental health problems.

ELIGIBILITY:
Inclusion Criteria:

* close to suicide victim or person who has mental health problems
* suicide victim or person with mental health problems was/is 45-60 years old
* the suicide happened more than 3 months and less than 5 years ago

Exclusion Criteria:

* not Dutch-speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
History of suicidal behaviour (presuicidal communication, method, intent) | baseline
Exposure to suicidal behavior | baseline
Sociodemographics | Baseline
Living situation | Baseline
Work situation | Baseline
Religion | Baseline
Interpersonal relationships (intimate, children, social contact, family) | Baseline
Financial problems | Baseline
Legal problems | Baseline
Life events | Baseline
Medical history | Baseline
Psychiatric history | Baseline
Psychiatric disorders | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kees van Heeringen, MD, PhD, Principal Investigator — University Ghent
Locations (1):
- Unit for Suicide Research, Ghent University, Ghent, Belgium